CLINICAL TRIAL: NCT01802671
Title: Cognitive Behavioural Treatment With Support on Communication and Information Technologies for the Management of Chronic Low Back Pain: A Randomized Clinical Trial
Brief Title: Efficacy Study of Cognitive Behavioural Treatment With Support on Communication and Information Technologies for the Management of Chronic Low Back Pain
Acronym: POETS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIS-PI12-02710
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Low Back Pain
Keywords: Low back pain; Cognitive behavioural treatment; internet; disability
MeSH Terms: conditions — Low Back Pain | interventions — Rehabilitation; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- cognitive behaviour therapy supported by ICT (Experimental): The patients of this group will receive the same interventions that the CBT group but will receive a reinforcements of the sessions' content through two different ways: a web tool named TEO (Emotional Therapy Online) and SMS that will send to the patients' mobile phone with reminders and reinforcements.
  Interventions: Other: Rehabilitation treatment and information; Behavioral: cognitive behavioural therapy (CBT); Behavioral: cognitive behaviour therapy supported by ICT
- Rehabilitation treatment and information (Active Comparator): Patients will receive the traditional rehabilitation treatment and information
  Interventions: Other: Rehabilitation treatment and information
- cognitive behavioural therapy (CBT) (Experimental): Patients will receive the same treatment in physical therapy than the control group and additionally they will receive CBT.
  Interventions: Other: Rehabilitation treatment and information; Behavioral: cognitive behavioural therapy (CBT)

INTERVENTIONS:
Other: Rehabilitation treatment and information — Patients will receive the traditional rehabilitation treatment (back school). This treatment will consist of a 4-session group therapy every week, with each session lasting 45 minutes. The content of the first session will be educational (ergonomics, pain demystification) and the other three will include physical therapy focused on stabilisation training: lower extremity stretching; finding the neutral spine position; spine stabiliser activation (transversus abdominis and multifidus); abdominal, spinal extensor and lower extremity strengthening; and proprioceptive control (stabilisation kinesitherapy)
Behavioral: cognitive behavioural therapy (CBT) — Patients will receive the same treatment in physical therapy than the control group and additionally they will receive CBT. The aim of the CBT intervention is to produce changes in the beliefs and behaviors about physical activity and avoidance of activity. The treatment's components are:
  * Psychoeducation to counteract the misconceptions about low back pain and to point on the relevance of maintaining an adequate level of activity.
  * Cognitive restructuring techniques
  * Behavioural therapy and activity pacing
  * Training on self-management pain techniques (mindfulness and relaxation). It is a 6-session group therapy, with one session per week. Each group will be composed by 6-8 participants. It will be considered as a patient who receives the treatment when the patient attends to the assessment sessions and to at least 4 out of 6 CBT sessions.
  Arms: cognitive behaviour therapy supported by ICT; cognitive behavioural therapy (CBT)
Behavioral: cognitive behaviour therapy supported by ICT — The patients of this group will receive the same interventions that the CBT group but will receive a reinforcements of the sessions' content through two different ways, both based on ICTs: a web tool named TEO (Emotional Therapy Online) specially designed to practicing the therapeutic strategies at home; and SMS that will send to the patients' mobile phone with reminders and reinforcements. The content of sessions will be related to the therapeutic components including on the CBT. Patients will access TEO from their home using a personal password. Besides TEO, messages will be sent through SMS three times per week during the treatment and once a week during the follow-up. The messages will consist on reminders to do the homework along with reinforcements of the working and effort made to improve their health.
  Arms: cognitive behaviour therapy supported by ICT

SUMMARY:
The objective of this study is to investigate the short- and long-term efficacy of a Cognitive Behavioural Treatment program for chronic low back pain supported by information and communication technologies

DETAILED DESCRIPTION:
Background: Psychological treatments have been successful in the treatment of chronic low back pain (CLBP). However the effect sizes are still modest and there is room for improvement. A way to progress in this line is enhancing treatment adherence and self-management by means of information and communication technologies (ICT). The objective of this study is to investigate the short- and long-term efficacy of a Cognitive Behavioural Treatment (CBT) group program for CLBP supported versus non-supported by ICTs. A secondary objective is to evaluate the influence of relevant variables in treatment response. Possible barriers in the implementation of CBT with and without ICT will be also investigated.

Methods: A randomized controlled trail with 180 CLBP patients recruited in specialized care will be conducted. Participants will be randomly assigned to three conditions: Control group (CG), Cognitive Behavioural program (CBT), and CBT supported by ICTs (CBT + ICT). Participants belonging to the three conditions will receive a conventional rehabilitation program (back school). The CBT group program will last six sessions. The CBT + ICT will use the Internet and SMS in order to practice the therapeutic strategies between sessions and in the follow-ups in their homes. Primary outcome variables are self-reported disability and pain intensity. Assessment will be carried out by blinded assessors in five moments: pre-treatment, post-treatment and 3-, 6-, and 12-month follow-up. The influence of catastrophizing, fear-avoidance beliefs, anxiety and depression in response to treatment in the primary outcomes will be also analysed.

Discussion This study will show data of the possible benefits of the use of ICTs in the improvement of CBT for the treatment of CLBP

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 65 years
* suffering low back pain for at least 6 months
* availability of mobile phone in order to get SMS
* access to computer with Internet connection in order to be able to use the CBT program supported by ICT

Exclusion Criteria:

* mental retardation
* not proficient in Spanish
* neurogenic claudication or neurologic deficit
* history of vertebral fracture, previous lumbar surgery
* vertebral infection
* spinal or nerve tumor
* severe mental disorder or substance abuse or dependence.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Disability: Change in the Roland-Morris Questionnaire | five assessment periods (pre-treatment, post-treatment, and three follow-ups at 3, 6 and 12 months).
  The Roland-Morris Questionnaire is one of the most widely used measures to assess disability in patients with low back pain, and it has shown good psychometrics properties (reliability and validity). The Spanish version of the RM will be completed by the patients. This questionnaire was designed to evaluate low back pain, with 24 statements that describe different daily activities that can be affected by low back pain. The participant has to select those statements that describe the limitations produced by low back pain.
Change in Pain measured by Numerical Rating Scale (NRS) | five assessment periods (pre-treatment, post-treatment, and three follow-ups at 3, 6 and 12 months).
  Pain: IMMPACT recommends the use of Numerical Rating Scales (NRS) as a core outcome measure of efficacy in clinical trials of chronic pain treatments. The scale is composed of 11 numbers ranging from 0 to 10 with 0 meaning 'No pain' and '10' meaning 'Pain as bad as you can imagine'. Two different scales will be used, one to assess low back pain and the other one to assess sciatica pain

SECONDARY OUTCOMES:
Change in Pain coping strategies | five assessment periods (pre-treatment, post-treatment, and three follow-ups at 3, 6 and 12 months).
  Pain coping strategies: The Coping Strategies Questionnaire (CSQ) assesses the frequency of several cognitive and behavioral strategies to cope with pain. Patients must select in a Likert-type scale how often they use each strategy. It comprises seven subscales, six for cognitive strategies (ignoring pain, reinterpretation of pain, diverting attention, coping self statements, catastrophizing, praying/hoping) and one subscale for behavioural strategies (activity level). This questionnaire has been validated in the Spanish population and has shown good psychometrics properties to the evaluation of patients with chronic musculoskeletal pain.
Change in Anxiety and Depression | five assessment periods (pre-treatment, post-treatment, and three follow-ups at 3, 6 and 12 months).
  Levels of anxiety and depression will be assessed by using the HADS questionnaire (Hospital Anxiety and Depression Score). This questionnaire is widely used in clinical practice. The HADS is a fourteen item scale where seven of the items are related to anxiety and the others seven are related to depression. The Spanish version has shown good internal consistency and external validity, as well as an adequate sensitivity in order to identify clinically significant depression.
Change in Fear-Avoidance Beliefs | five assessment periods (pre-treatment, post-treatment, and three follow-ups at 3, 6 and 12 months).
  The Fear-Avoidance Beliefs Questionnaire (FABQ) will be used to measure this domain. Is a scale composed by sixteen items developed to assess patients' beliefs and attitudes about the causes and consequences of their low back pain. Participants rate their agreement with each statement on a 7- point Likert scale (0 = completely disagree, 6 = completely agree). The FABQ consists of 2 subscales. The first sub-scale is the Physical Activity subscale (FABQpa), is composed by seven items, and assesses the effects of physical activities over pain. The second subscale is the Work subscale (FABQw) composed by four items, and it assesses the way that work activities can affect pain. The Spanish version has shown excellent psychometrics properties.
Change in Catastrophizing | five assessment periods (pre-treatment, post-treatment, and three follow-ups at 3, 6 and 12 months).
  The Pain Catastrophizing Scale (PCS) assesses the tendency to consider pain as a threat with exaggerated negative consequence to the patient. It is a 13-item self-report scale, each item evaluate the pain experience, as an example: "I become afraid that the pain will get worse". Participants assess the frequency that these ideas appears, on a likert-type scale ranging from 0 to 4 being 0 "not at all" and 4 "all the time". The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness. A high score on the total PCS score indicates a high level of catastrophizing. The Spanish version of PCS has demonstrated adequate psychometrics properties.
Change in Quality of life assessed by the SF-12 questionnaire | five assessment periods (pre-treatment, post-treatment, and three follow-ups at 3, 6 and 12 months).
  The SF-12 is the brief version of the 36-item Short Form Health Survey (SF-36). The SF-12 contains items that measure each of the eight concepts included in the SF-36, namely physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being). The SF-12 contains six-point scales were patients evaluated the frequency and intensity of each statement during the past month.

OTHER OUTCOMES:
Satisfaction with the treatment: The Spanish adaptation of Borkovec and Nau questionnaire | 12 months
  Satisfaction with the treatment: The Spanish adaptation of Borkovec and Nau questionnaire (1972) will be used. Participants have to respond in an eleven-point scale (0 to 10) several questions about their opinion over the received treatment (for example, how logic was the treatment for them; if they are satisfied; if the treatment was useful; if they would recommend the treatment to other people). Clinicians will also be assessed with an adapted version of the questionnaire regarding satisfaction with the treatment program.
Analysis of the barriers for the use of cognitive behavioral therapy and communication and information technologies in chronic low back pain treatment: | 12 months
  Analysis of the barriers for the use of cognitive behavioral therapy and communication and information technologies in chronic low back pain treatment: This analysis includes 3 groups of patients, resulting from the three experimental conditions, compound of 8 patients each, selected by a balanced randomization to assure variability in gender, age, educational levels and level's use of information and communication technologies. We will apply a focus group strategy and it will be accomplished at the end of the therapy. The focus groups will be recorded and analyzed with qualitative analysis methodology. The clinic staff's opinion will be obtained on ad-hoc questionnaires and filled in by the clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Domenech, Md PhD, Orthopedic Surgery, Principal Investigator — Hospital Arnau de Vilanova, Valencia
Locations (1):
- Hospital Arnau de Vilanova, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Domenech J, Banos R, Penalver L, Garcia-Palacios A, Herrero R, Ezzedine A, Martinez-Diaz M, Ballester J, Horta J, Botella C. Design considerations of a randomized clinical trial on a cognitive behavioural intervention using communication and information technologies for managing chronic low back pain. BMC Musculoskelet Disord. 2013 Apr 22;14:142. doi: 10.1186/1471-2474-14-142. PMID 23607895